CLINICAL TRIAL: NCT04351568
Title: Professional and Ethical Challenges of Social Media Usage in Providing Healthcare Services; During the Period of 19 Covid Pandemics
Brief Title: Professional and Ethical Challenges of Social Media Usage in Providing Healthcare Services During the Period of 19 Covid Pandemics;
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Esmael Ebrahem, faculty of medicine assuit university, Assiut University
Other Study IDs: 2020A20
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Evaluating the Effect of Social Media Usage in Providing Healthcare Services During the Period of 19 Covid Pandemics

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- medical personel
  Interventions: Other: quesionnair
- non medical personel
  Interventions: Other: quesionnair

INTERVENTIONS:
Other: quesionnair — questionnair about Emerging Legal and Ehical Disputes Over Patient Confidentiality

SUMMARY:
integrating social media into medicine has obvious potential to improve patient care and trust in the profession, in part by meeting patients "where they are," i.e., online, at the same time carries a greater risk in terms of legal, ethical, and professional aspects. Therefore, physicians and medical students using social media should pay attention to the ethical sensitivity in their relationships with patients .it also raises a number of ethical issues including protecting patient and physician privacy; setting appropriate online boundaries; and delineating personal and professional identities among others during covid 19 pandemics

ELIGIBILITY:
Inclusion Criteria:

1. adult aged 18 years to 60 years
2. medical personel graduated from egyptian faculty of medicine.
3. non medical personel live in egypt

Exclusion Criteria:

1. personel less than 18 years old .
2. medical personel not graduated from egyptian faculty of medicine.
3. non medical personel live outside egypt

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: medical and non medical personel
Sampling Method: Probability Sample
Enrollment: 874 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
to evaluate the effect of social media usage in medical practice during covid 19 epidemic | 3 months
  to evaluate the effect of social media usage in medical practice during covid 19 epidemic

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut, Asyut, Egypt